CLINICAL TRIAL: NCT02260986
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Demonstrate the Efficacy and Long-Term Safety of Dupilumab in Adult Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study to Assess the Efficacy and Long-term Safety of Dupilumab (REGN668/SAR231893) in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: CHRONOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1224
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo qw (Experimental): Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection weekly (qw) from Week 1 to Week 51.
  Interventions: Drug: Placebo (for Dupilumab); Other: Topical Corticosteroid (TCS)
- Dupilumab 300 mg q2w (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab every 2 weeks (q2w) from Week 1 to Week 51. During weeks in which Dupilumab was not administered, participants received placebo.
  Interventions: Drug: Dupilumab; Drug: Placebo (for Dupilumab); Other: Topical Corticosteroid (TCS)
- Dupilumab 300 mg qw (Experimental): Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab qw from Week 1 to Week 51.
  Interventions: Drug: Dupilumab; Other: Topical Corticosteroid (TCS)

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection in the different quadrants of the abdomen (avoiding navel and waist areas) and upper thighs
  Other Names: REGN668; SAR231893; Dupixent
  Arms: Dupilumab 300 mg q2w; Dupilumab 300 mg qw
Drug: Placebo (for Dupilumab) — Subcutaneous injection in the different quadrants of the abdomen (avoiding navel and waist areas) and upper thighs
  Arms: Dupilumab 300 mg q2w; Placebo qw
Other: Topical Corticosteroid (TCS) — All participants were required to treatment with a (TCS) using a standardized regimen. It was recommended that participants use triamcinolone acetonide 0.1% cream or fluocinolone acetonide 0.025% ointment for medium potency, and hydrocortisone 1% cream for low potency.

SUMMARY:
The primary objective of the study was to demonstrate the efficacy of Dupilumab administered concomitantly with topical corticosteroid (TCS) through Week 16 in adult participants with moderate-to-severe atopic dermatitis (AD) compared to placebo administered concomitantly with TCS.

ELIGIBILITY:
Key Inclusion Criteria:

1. Chronic AD that had been present for at least 3 years before the screening visit;
2. Documented recent history (within 6 months before the screening visit) of inadequate response to a sufficient course of out-patient treatment with topical AD medication(s).

Key Exclusion Criteria:

1. Participation in a prior Dupilumab clinical trial;
2. Important side effects of topical medication (e.g. intolerance to treatment, hypersensitivity reactions, significant skin atrophy, systemic effects), as assessed by the investigator or treating physician;
3. Having used any of the following treatments within 4 weeks before the baseline visit, or any condition that, in the opinion of the investigator, was likely to require such treatment(s) during the first 2 weeks of study treatment:

   1. Immunosuppressive/immunomodulating drugs (e.g, systemic steroids, cyclosporine, mycophenolate-mofetil, Janus kinase inhibitors, interferon-gamma [IFN-γ], azathioprine, methotrexate, etc.);
   2. Phototherapy for AD;
4. Treatment with a live (attenuated) vaccine within 12 weeks before the baseline visit;
5. History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening;
6. Positive hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody at the screening visit;
7. Active or acute infection requiring systemic treatment within 2 weeks before baseline visit;
8. Known or suspected history of immunosuppression;
9. Pregnant or breastfeeding women, or planning to become pregnant or breastfeed during the participant's participation in this study.

Note: The eligibility criteria listed above is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial therefore not all inclusion/ exclusion criteria are listed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (148):
- United States (50):
  - Phoenix, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Encinitas, California
  - Oceanside, California
  - Palmdale, California
  - San Diego, California
  - New Haven, Connecticut
  - Trumbull, Connecticut
  - Edgewater, Florida
  - Lake Worth, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - West Dundee, Illinois
  - Carmel, Indiana
  - New Albany, Indiana
  - Rockville, Maryland
  - Ann Arbor, Michigan
  - Bay City, Michigan
  - Edina, Minnesota
  - Fridley, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Henderson, Nevada
  - Verona, New Jersey
  - Albuquerque, New Mexico
  - Corning, New York
  - New York, New York
  - Smithtown, New York
  - Stony Brook, New York
  - Cincinnati, Ohio
  - Norman, Oklahoma
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Exton, Pennsylvania
  - Hazleton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - West Jordan, Utah
  - South Burlington, Vermont
  - Henrico, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Spokane, Washington
- Australia (6):
  - Phillip, Australian Capital Territory
  - Kogarah, New South Wales
  - Benowa, Queensland
  - Dulwich, Queensland
  - Hectorville, South Australia
  - Carlton, Victoria
- Canada (16):
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Ajax, Ontario
  - Barrie, Ontario
  - Hamilton, Ontario
  - Markham, Ontario
  - North Bay, Ontario
  - Oakville, Ontario
  - Ottawa, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Drummondville, Quebec
  - Québec
- Czechia (5):
  - Hradec Králové
  - Náchod
  - Prague
  - Svitavy
  - Ústí nad Labem
- Hungary (4):
  - Orosháza, Bekes County
  - Szolnok, Jász-Nagykun-Szolnok
  - Veszprém, Veszprém megye
  - Budapest
- Italy (7):
  - Ancona
  - Bologna
  - Brescia
  - Novara
  - Pavia
  - Perugia
  - Roma
- Japan (17):
  - Kitakyushu, Fukuoka
  - Amagasaki, Hyôgo
  - Yokohama, Kanagawa
  - Kamimashiki-gun, Kumamoto
  - Saitama-shi, Saitama
  - Yaizu, Shizuoka
  - Koto-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Adachi-ku, Tôkyô
  - Chiyoda-ku, Tôkyô
  - Nakano, Tôkyô
  - Nerima-ku, Tôkyô
  - Shibuya-ku, Tôkyô
  - Shinagawa-ku, Tôkyô
  - Shinjuku-ku, Tôkyô
  - Suginami-ku, Tôkyô
  - Fukuoka
- Netherlands (5):
  - Breda, North Brabant
  - Amsterdam, North Holland
  - Rotterdam, South Holland
  - Groningen
  - Utrecht
- New Zealand (2):
  - Dunedin, South Island
  - Auckland
- Poland (14):
  - Poznan, Greater Poland Voivodeship
  - Krakow, Lesser Poland Voivodeship
  - Wroclaw, Lower Silesian Voivodeship
  - Lublin, Lublin Voivodeship
  - Warsaw, Masovian Voivodeship
  - Strzelce Opolskie, Opole Voivodeship
  - Iwonicz-Zdrój, Podkarpackie Voivodeship
  - Bialystok, Podlaskie Voivodeship
  - Gdansk, Pomeranian Voivodeship
  - Katowice, Silesian Voivodeship
  - Szczecin, West Pomeranian Voivodeship
  - Gdynia
  - Lodz, Łódź Voivodeship
  - Skarżysko-Kamienna, Świętokrzyskie Voivodeship
- Romania (5):
  - Brasov, Brașov County
  - Bucharest, București
  - Cluj-Napoca, Cluj
  - Craiova, Dolj
  - Târgu Mureş, Mureș County
- South Korea (5):
  - Bucheon-si, Gyeonggido
  - Suwon, Gyeonggido
  - Seoul, Seoul Teugbyeolsi
  - Seodaemun-gu
  - Uijeongbu-si
- Spain (3):
  - Barcelona, Catalonia
  - Alicante
  - Madrid
- United Kingdom (9):
  - Dundee, Angus
  - Edgbaston, Birmingham
  - Glasgow, Glasgow City
  - Sidcup, Kent
  - Northwood, Middlesex
  - Liverpool
  - Manchester
  - Reading
  - Salford

REFERENCES:
- [Derived] Simpson EL, Bissonnette R, Deleuran M, Nakahara T, Galus R, de Bruin-Weller M, Coleman A, van Spall M, Chen Z, Avetisova E, Bastian M, Khokhar FA. Dupilumab Treatment Up to 5 Years Shows No Clinically Meaningful Changes in Laboratory Parameters in Adults with Moderate-to-Severe Atopic Dermatitis. Adv Ther. 2026 Jan 21. doi: 10.1007/s12325-025-03458-3. Online ahead of print. PMID 41563707
- [Derived] Yosipovitch G, Kim BS, Koo JY, Chen Z, Wiggins S, Zahn J, Sugerman P, Haddad EB, Cyr SL. Dupilumab Reduces Pruritus in Clinically Distinct Dermatologic Diseases: Data from Clinical Trials on Atopic Dermatitis, Prurigo Nodularis, and Chronic Spontaneous Urticaria. Dermatol Ther (Heidelb). 2025 Nov 22. doi: 10.1007/s13555-025-01596-8. Online ahead of print. PMID 41272364
- [Derived] Wiseman M, Benvenuto M, Stromkjaer L, Paludan-Muller A, Ryttig L, Petersen AS, Wollenberg A. Cost-Per-Responder Analysis for Tralokinumab and Dupilumab in Combination with Topical Corticosteroids in Patients with Moderate-To-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Oct 16. doi: 10.1007/s13555-025-01565-1. Online ahead of print. PMID 41102518
- [Derived] Langley RG, Gherardi G, Coleman A, Ardeleanu M, Rodriguez-Marco A, Levy S, Bansal A, Chen Z, Rossi AB, Shumel B, Khokhar FA. The Safety Data of Dupilumab for the Treatment of Moderate-to-Severe Atopic Dermatitis in Infants, Children, Adolescents, and Adults. Am J Clin Dermatol. 2025 Nov;26(6):981-1002. doi: 10.1007/s40257-025-00952-w. Epub 2025 Sep 24. PMID 40993471
- [Derived] Stander S, Yosipovitch G, Kim BS, Steinhoff M, Armstrong A, Legat FJ, Kabashima K, Nakahara T, Igarashi A, Praestgaard AH, Nguyen TV, Bastian M. Optimal Itch Response in Adults Treated with Dupilumab for Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Nov;15(11):3437-3446. doi: 10.1007/s13555-025-01519-7. Epub 2025 Sep 19. PMID 40971025
- [Derived] Stander S, Yosipovitch G, Simpson EL, Kim BS, Kabashima K, Thaci D, Metz M, Chen Z, Hagen S, Bastian M. Onset and Long-Term Maintenance of Optimal Itch Response in Adult Patients with Moderate-to-Severe Atopic Dermatitis Treated with Dupilumab: Post Hoc Analysis from Two Phase 3 Trials. Adv Ther. 2025 Apr;42(4):1800-1810. doi: 10.1007/s12325-025-03124-8. Epub 2025 Feb 19. PMID 39969783
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Silverberg JI, Lynde CW, Abuabara K, Patruno C, de Benedetto A, Zhang H, Thomas RB, Bego-Le-Bagousse G, Khokhar FA, Vakil J, Marco AR, Levit NA. Efficacy and Safety of Dupilumab Maintained in Adults >/= 60 Years of Age with Moderate-to-Severe Atopic Dermatitis: Analysis of Pooled Data from Four Randomized Clinical Trials. Am J Clin Dermatol. 2023 May;24(3):469-483. doi: 10.1007/s40257-022-00754-4. Epub 2023 Feb 20. PMID 36808602
- [Derived] Paller AS, Silverberg JI, Cork MJ, Guttman-Yassky E, Lockshin B, Irvine AD, Kim MB, Kabashima K, Chen Z, Lu Y, Bansal A, Rossi AB, Shabbir A. Efficacy and Safety of Dupilumab in Patients With Erythrodermic Atopic Dermatitis: A Post Hoc Analysis of 6 Randomized Clinical Trials. JAMA Dermatol. 2023 Mar 1;159(3):255-266. doi: 10.1001/jamadermatol.2022.6192. PMID 36723913
- [Derived] Wechsler ME, Klion AD, Paggiaro P, Nair P, Staumont-Salle D, Radwan A, Johnson RR, Kapoor U, Khokhar FA, Daizadeh N, Chen Z, Laws E, Ortiz B, Jacob-Nara JA, Mannent LP, Rowe PJ, Deniz Y. Effect of Dupilumab on Blood Eosinophil Counts in Patients With Asthma, Chronic Rhinosinusitis With Nasal Polyps, Atopic Dermatitis, or Eosinophilic Esophagitis. J Allergy Clin Immunol Pract. 2022 Oct;10(10):2695-2709. doi: 10.1016/j.jaip.2022.05.019. Epub 2022 May 28. PMID 35636689
- [Derived] Blauvelt A, de Bruin-Weller M, Simpson EL, Chen Z, Ardeleanu M, Rossi AB. Consistency of Response to Dupilumab in Adults with Moderate-to-Severe Atopic Dermatitis Over 1 Year. Dermatol Ther (Heidelb). 2022 Jan;12(1):9-13. doi: 10.1007/s13555-021-00657-y. Epub 2022 Jan 7. PMID 34994968
- [Derived] Blauvelt A, de Bruin-Weller M, Simpson EL, Chen Z, Zhang A, Shumel B. Dupilumab with Topical Corticosteroids Provides Rapid and Sustained Improvement in Adults with Moderate-to-Severe Atopic Dermatitis Across Anatomic Regions Over 52 Weeks. Dermatol Ther (Heidelb). 2022 Jan;12(1):223-231. doi: 10.1007/s13555-021-00638-1. Epub 2021 Nov 22. PMID 34806137
- [Derived] Griffiths C, de Bruin-Weller M, Deleuran M, Fargnoli MC, Staumont-Salle D, Hong CH, Sanchez-Carazo J, Foley P, Seo SJ, Msihid J, Chen Z, Cyr SL, Rossi AB. Dupilumab in Adults with Moderate-to-Severe Atopic Dermatitis and Prior Use of Systemic Non-Steroidal Immunosuppressants: Analysis of Four Phase 3 Trials. Dermatol Ther (Heidelb). 2021 Aug;11(4):1357-1372. doi: 10.1007/s13555-021-00558-0. Epub 2021 Jun 18. PMID 34142350
- [Derived] Hamilton JD, Harel S, Swanson BN, Brian W, Chen Z, Rice MS, Amin N, Ardeleanu M, Radin A, Shumel B, Ruddy M, Patel N, Pirozzi G, Mannent L, Graham NMH. Dupilumab suppresses type 2 inflammatory biomarkers across multiple atopic, allergic diseases. Clin Exp Allergy. 2021 Jul;51(7):915-931. doi: 10.1111/cea.13954. Epub 2021 Jun 26. PMID 34037993
- [Derived] Wu JJ, Spelman L, Tan JL, Etoh T, Zhang H, Shumel B, Rossi AB. Dupilumab Maintains Long-Term Disease Control in Adults with Moderate-to-Severe Atopic Dermatitis as Measured by Well-Controlled Weeks: Results From the LIBERTY AD CHRONOS Clinical Trial. Dermatol Ther (Heidelb). 2021 Apr;11(2):327-330. doi: 10.1007/s13555-021-00487-y. Epub 2021 Jan 28. No abstract available. PMID 33511576
- [Derived] Boguniewicz M, Beck LA, Sher L, Guttman-Yassky E, Thaci D, Blauvelt A, Worm M, Corren J, Soong W, Lio P, Rossi AB, Lu Y, Chao J, Eckert L, Gadkari A, Hultsch T, Ruddy M, Mannent LP, Graham NMH, Pirozzi G, Chen Z, Ardeleanu M. Dupilumab Improves Asthma and Sinonasal Outcomes in Adults with Moderate to Severe Atopic Dermatitis. J Allergy Clin Immunol Pract. 2021 Mar;9(3):1212-1223.e6. doi: 10.1016/j.jaip.2020.12.059. Epub 2021 Jan 13. PMID 33453450
- [Derived] Silverberg JI, Simpson EL, Guttman-Yassky E, Cork MJ, de Bruin-Weller M, Yosipovitch G, Eckert L, Chen Z, Ardeleanu M, Shumel B, Hultsch T, Rossi AB, Hamilton JD, Orengo JM, Ruddy M, Graham NMH, Pirozzi G, Gadkari A. Dupilumab Significantly Modulates Pain and Discomfort in Patients With Atopic Dermatitis: A Post Hoc Analysis of 5 Randomized Clinical Trials. Dermatitis. 2021 Oct 1;32(1S):S81-S91. doi: 10.1097/DER.0000000000000698. PMID 33165005
- [Derived] Weyne J, Blauvelt A, de Bruin-Weller M, Prens E, Asbell P, Sierka D, Chen Z, Shumel B. Patient-Reported Ocular Disorders and Symptoms in Adults with Moderate-to-Severe Atopic Dermatitis: Screening and Baseline Survey Data from a Clinical Trial. Dermatol Ther (Heidelb). 2020 Dec;10(6):1415-1421. doi: 10.1007/s13555-020-00456-x. Epub 2020 Oct 12. PMID 33047298
- [Derived] Katoh N, Kataoka Y, Saeki H, Hide M, Kabashima K, Etoh T, Igarashi A, Imafuku S, Kawashima M, Ohtsuki M, Fujita H, Arima K, Takagi H, Chen Z, Shumel B, Ardeleanu M. Efficacy and safety of dupilumab in Japanese adults with moderate-to-severe atopic dermatitis: a subanalysis of three clinical trials. Br J Dermatol. 2020 Jul;183(1):39-51. doi: 10.1111/bjd.18565. Epub 2019 Nov 28. PMID 31564057
- [Derived] Alexis AF, Rendon M, Silverberg JI, Pariser DM, Lockshin B, Griffiths CE, Weisman J, Wollenberg A, Chen Z, Davis JD, Li M, Eckert L, Gadkari A, Shumel B, Rossi AB, Graham NM, Ardeleanu M. Efficacy of Dupilumab in Different Racial Subgroups of Adults With Moderate-to-Severe Atopic Dermatitis in Three Randomized, Placebo-Controlled Phase 3 Trials. J Drugs Dermatol. 2019 Aug 1;18(8):804-813. PMID 31424712
- [Derived] Wollenberg A, Beck LA, Blauvelt A, Simpson EL, Chen Z, Chen Q, Shumel B, Khokhar FA, Hultsch T, Rizova E, Rossi AB, Graham NMH, Pirozzi G, Lu Y, Ardeleanu M. Laboratory safety of dupilumab in moderate-to-severe atopic dermatitis: results from three phase III trials (LIBERTY AD SOLO 1, LIBERTY AD SOLO 2, LIBERTY AD CHRONOS). Br J Dermatol. 2020 May;182(5):1120-1135. doi: 10.1111/bjd.18434. Epub 2019 Dec 1. PMID 31407311
- [Derived] Eichenfield LF, Bieber T, Beck LA, Simpson EL, Thaci D, de Bruin-Weller M, Deleuran M, Silverberg JI, Ferrandiz C, Folster-Holst R, Chen Z, Graham NMH, Pirozzi G, Akinlade B, Yancopoulos GD, Ardeleanu M. Infections in Dupilumab Clinical Trials in Atopic Dermatitis: A Comprehensive Pooled Analysis. Am J Clin Dermatol. 2019 Jun;20(3):443-456. doi: 10.1007/s40257-019-00445-7. PMID 31066001
- [Derived] Blauvelt A, de Bruin-Weller M, Gooderham M, Cather JC, Weisman J, Pariser D, Simpson EL, Papp KA, Hong HC, Rubel D, Foley P, Prens E, Griffiths CEM, Etoh T, Pinto PH, Pujol RM, Szepietowski JC, Ettler K, Kemeny L, Zhu X, Akinlade B, Hultsch T, Mastey V, Gadkari A, Eckert L, Amin N, Graham NMH, Pirozzi G, Stahl N, Yancopoulos GD, Shumel B. Long-term management of moderate-to-severe atopic dermatitis with dupilumab and concomitant topical corticosteroids (LIBERTY AD CHRONOS): a 1-year, randomised, double-blinded, placebo-controlled, phase 3 trial. Lancet. 2017 Jun 10;389(10086):2287-2303. doi: 10.1016/S0140-6736(17)31191-1. Epub 2017 May 4. PMID 28478972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 14 countries between 16 Sep 2014 and 19 Oct 2016. A total of 957 participants were screened in the study.
Pre-assignment Details: Out of 957 participants, 740 participants were randomized and treated in the study. Participants were randomized in 3:1:3 ratio to receive Dupilumab 300 mg once weekly (qw) or Dupilumab 300 mg every 2 weeks (q2w) or placebo (for Dupilumab) qw.
Groups:
- Placebo qw: Two subcutaneous injections of Placebo (for Dupilumab) as a loading dose on Day 1 followed by a single injection qw from Week 1 to Week 51.
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 51. During weeks in which Dupilumab was not administered, participants received placebo.
Period: Overall Study
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Started | 315 | 106 | 319
Safety Population | 315 | 110 (4 participants from Dupilumab 300 mg qw arm analyzed in Dupilumab 300 mg q2w arm) | 315 (4 participants received fewer injections of Dupilumab 300 mg (analyzed in Dupilumab 300 mg q2w arm))
Completed | 225 | 93 | 278
Not Completed | 90 | 13 | 41
Not completed — Adverse Event | 24 | 0 | 11
Not completed — Lack of Efficacy | 27 | 3 | 0
Not completed — Protocol Violation | 14 | 5 | 16
Not completed — Car accident | 0 | 0 | 1
Not completed — Withdrawal by Subject | 17 | 4 | 9
Not completed — Incorrect randomization | 0 | 1 | 0
Not completed — Lack of investigation product supply | 2 | 0 | 1
Not completed — Lost to Follow-up | 4 | 0 | 3
Not completed — Pregnancy | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw | Total
Number analyzed (Participants) | 315 | 106 | 319 | 740
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (13.01) | 39.6 (13.98) | 36.9 (13.67) | 37.1 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 44 | 128 | 294
  Male | 193 | 62 | 191 | 446
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 5 | 17
  Not Hispanic or Latino | 299 | 103 | 309 | 711
  Unknown or Not Reported | 6 | 1 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 83 | 29 | 89 | 201
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 2 | 13 | 34
  White | 208 | 74 | 208 | 490
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 9 | 15
Region of Enrollment [Number; unit: participants]
  Romania | 2 | 0 | 2 | 4
  Hungary | 11 | 5 | 11 | 27
  United States | 61 | 19 | 59 | 139
  Japan | 54 | 16 | 47 | 117
  United Kingdom | 17 | 4 | 15 | 36
  Spain | 4 | 2 | 4 | 10
  New Zealand | 1 | 1 | 3 | 5
  Canada | 47 | 17 | 51 | 115
  Czech Republic | 7 | 7 | 6 | 20
  Netherlands | 17 | 7 | 19 | 43
  Korea, Republic of | 8 | 4 | 14 | 26
  Poland | 63 | 17 | 64 | 144
  Italy | 5 | 1 | 7 | 13
  Australia | 18 | 6 | 17 | 41
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
  units on a scale | 32.6 (12.93) | 33.6 (13.30) | 32.1 (12.76) | 32.5 (12.90)
Investigator Global Assessment (IGA) Score [Mean (Standard Deviation); unit: units on a scale] — IGA was an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response was an IGA score of 0 (clear) or 1 (almost clear).
  units on a scale | 3.5 (0.50) | 3.5 (0.50) | 3.5 (0.50) | 3.5 (0.50)
Weekly Peak Averaged Pruritus Numeric Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS was an assessment tool that was used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at worst moment during previous 24 hours (for maximum itch intensity on a scale of 0-10 [0=no itch;10=worst itch imaginable]).
  units on a scale | 7.3 (1.84) | 7.4 (1.66) | 7.1 (1.90) | 7.3 (1.84)
Body Surface Area (BSA) Involvement with Atopic Dermatitis [Mean (Standard Deviation); unit: Percentage of body surface area] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  Percentage of body surface area | 56.9 (21.69) | 59.5 (20.84) | 54.1 (21.76) | 56.1 (21.66)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD is a clinical tool for assessing the severity of atopic dermatitis developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Population: Number of participants analyzed = participants with available data for this baseline parameter.
  units on a scale
    number analyzed (Participants) | 313 | 105 | 316 | 734
    (all) | 66.0 (13.53) | 69.3 (15.24) | 65.9 (13.63) | 66.4 (13.86)
Dermatology Life Quality Index (DLQI) Total Score [Mean (Standard Deviation); unit: units on a scale] — DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL.
  units on a scale | 14.7 (7.37) | 14.5 (7.31) | 14.4 (7.17) | 14.5 (7.27)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: units on a scale] — The POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). Population: Number of participants analyzed = participants with available data for this baseline parameter.
  units on a scale
    number analyzed (Participants) | 314 | 106 | 319 | 739
    (all) | 20.0 (5.99) | 20.3 (5.68) | 20.1 (6.05) | 20.1 (5.95)
Global Individual Signs Score (GISS) [Mean (Standard Deviation); unit: units on a scale] — Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0 = none, 1 = mild, 2 = moderate and 3 = severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
  units on a scale | 8.7 (1.84) | 8.9 (2.04) | 8.9 (1.80) | 8.8 (1.85)
Total Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
  units on a scale | 12.6 (8.06) | 12.9 (7.73) | 12.8 (8.01) | 12.7 (7.98)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Reduction From Baseline of ≥2 Points at Week 16
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score "0" or "1" and a reduction from baseline of ≥2 points at Week 16 were reported.
Time Frame: Baseline to Week 16
Population: All efficacy analyses were performed on the Full Analysis Set (FAS), which included all randomized participants. Efficacy analyses were based on the treatment allocated by interactive voice response system/ interactive web response system (IVRS/IWRS) at randomization (as randomized).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percentage of participants | 12.4 | 38.7 | 39.2
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 16 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 26.3, 95% CI 2-sided [16.34 to 36.26] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 26.8, 95% CI 2-sided [20.33 to 33.28] — Dupilumab 300 mg qw v Placebo

2. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) at Week 16
Description: The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 16.
Time Frame: Baseline to Week 16
Population: All efficacy analyses were performed on the FAS, which included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized).
Measure: Number; unit: percentage of participants
Groups:
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 51.
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percentage of participants | 23.2 | 68.9 | 63.9
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.025 level for both comparisons; Test type: Superiority — Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment use were set to missing and participants with missing EASI score at Week 16 were considered as non-responders; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 45.7, 95% CI 2-sided [35.72 to 55.66] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; A hierarchical testing procedure was used to control type I error and handle multiple secondary endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when previous endpoint was statistically significant at 0.025 level for both comparisons; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 40.8, 95% CI 2-sided [33.74 to 47.81] — Dupilumab 300 mg qw v Placebo

3. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported.
Time Frame: Baseline to Week 16
Population: All efficacy analyses were performed on the FAS, which included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized). Here, number of participants analyzed = participants with baseline peak pruritus NRS score ≥4.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 299 | 102 | 295
percentage of participants | 19.7 | 58.8 | 50.8
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment use were set to missing and participants with missing peak NRS at Week 16 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 39.1, 95% CI 2-sided [28.53 to 49.65] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 31.1, 95% CI 2-sided [23.84 to 38.39] — Dupilumab 300 mg qw v Placebo

4. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥3 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥3 points from baseline in weekly average of peak daily pruritus NRS score at Week 16 were reported.
Time Frame: Baseline to Week 16
Population: All efficacy analyses were performed on the FAS, which included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized). Here, number of participants analyzed = participants with baseline peak pruritus NRS score ≥3.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 306 | 105 | 309
percentage of participants | 27.8 | 65.7 | 62.5
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 37.9, 95% CI 2-sided [27.56 to 48.31] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 34.7, 95% CI 2-sided [27.31 to 42.05] — Dupilumab 300 mg qw v Placebo

5. Secondary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of "0" or "1" and Reduction From Baseline of ≥2 Points at Week 52
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of "0" or "1" and a reduction from baseline of ≥2 points at Week 52 were reported.
Time Frame: Baseline to Week 52
Population: All efficacy analyses were performed on the FAS, which included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized). Here, number of participants analyzed = participants with available data for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
percentage of participants | 12.5 | 36.0 | 40.0
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 52 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 23.5, 95% CI 2-sided [12.72 to 34.19] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.5, 95% CI 2-sided [20.42 to 34.58] — Dupilumab 300 mg qw v Placebo

6. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-75 (EASI-75) (≥75% Improvement From Baseline) at Week 52
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved ≥75% overall improvement in EASI score from baseline to Week 52.
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
percentage of participants | 21.6 | 65.2 | 64.1
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment use were set to missing and participants with missing EASI score at Week 52 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 43.6, 95% CI 2-sided [32.50 to 54.65] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 42.5, 95% CI 2-sided [34.91 to 50.06] — Dupilumab 300 mg qw v Placebo

7. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percent change | -30.3 (2.36) | -56.6 (3.95) | -57.1 (2.11)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using ANCOVA model with baseline measurements as covariate and the treatment, region and baseline IGA strata as fixed factors; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; Least square (LS) mean difference = -26.2, 95% CI 2-sided [-35.04 to -17.43] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -26.8, 95% CI 2-sided [-32.83 to -20.73] — Dupilumab 300 mg qw v Placebo

8. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 52
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 52 were reported.
Time Frame: Baseline to Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 249 | 86 | 249
percentage of participants | 12.9 | 51.2 | 39.0
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 52 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 38.3, 95% CI 2-sided [26.96 to 49.66] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 26.1, 95% CI 2-sided [18.76 to 33.45] — Dupilumab 300 mg qw v Placebo

9. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥3 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 52
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥3 points from baseline in weekly average of peak daily pruritus NRS score at Week 52 were reported.
Time Frame: Baseline to Week 52
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 256 | 88 | 261
percentage of participants | 15.6 | 55.7 | 42.9
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 40.1, 95% CI 2-sided [28.76 to 51.35] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.3, 95% CI 2-sided [19.81 to 34.76] — Dupilumab 300 mg qw v Placebo

10. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 24
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 24 were reported.
Time Frame: Baseline to Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 299 | 102 | 295
percentage of participants | 16.1 | 53.9 | 43.7
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 24 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 37.9, 95% CI 2-sided [27.34 to 48.40] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 27.7, 95% CI 2-sided [20.65 to 34.70] — Dupilumab 300 mg qw v Placebo

11. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 4
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 4 were reported.
Time Frame: Baseline to Week 4
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 299 | 102 | 295
percentage of participants | 16.4 | 37.3 | 27.1
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 4 were considered as non-responders; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 20.9, 95% CI 2-sided [10.59 to 31.15] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 10.7, 95% CI 2-sided [4.15 to 17.31] — Dupilumab 300 mg qw v Placebo

12. Secondary Outcome: Percentage of Participants With Improvement (Reduction ≥4 Points) of Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 2
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Participants achieving a reduction of ≥4 points from baseline in weekly average of peak daily pruritus NRS score at Week 2 were reported.
Time Frame: Baseline to Week 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 299 | 102 | 295
percentage of participants | 8.0 | 17.6 | 13.6
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region and baseline disease severity (IGA baseline values: IGA=3 vs IGA=4). Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 2 were considered as non-responders; Test type: Superiority; p = 0.0062, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 9.6, 95% CI 2-sided [1.61 to 17.63] — Dupilumab 300 mg q2w v Placebo
Statistical Analysis 2: Comparison: Placebo qw vs Dupilumab 300 mg qw; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0344, Cochran-Mantel-Haenszel — Threshold for significance at 0.025 level; difference in percentages = 5.5, 95% CI 2-sided [0.56 to 10.51] — Dupilumab 300 mg qw v Placebo

13. Secondary Outcome: Change From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 16
Description: as for outcome 7
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
units on a scale | -2.36 (0.138) | -4.17 (0.207) | -4.27 (0.126)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -1.81, 95% CI 2-sided [-2.297 to -1.322] — Dupilumab 300 mg q2w v Placebo

14. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score to Week 16
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 188 | 92 | 269
percent change | -48.4 (3.82) | -80.5 (6.34) | -81.5 (5.78)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -32.1, 95% CI 2-sided [-46.37 to -17.82] — Dupilumab 300 mg q2w v Placebo

15. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Atopic Dermatitis to Week 16
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of BSA
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
Percentage of BSA | -22.01 (1.158) | -40.39 (1.844) | -39.58 (1.065)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -18.38, 95% CI 2-sided [-22.583 to -14.187] — Dupilumab 300 mg q2w v Placebo

16. Secondary Outcome: Percent Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Score to Week 16
Description: SCORAD was a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percent change | -36.2 (1.66) | -63.9 (2.52) | -65.9 (1.49)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -27.7, 95% CI 2-sided [-33.46 to -21.9] — Dupilumab 300 mg q2w v Placebo

17. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 16
Description: The DLQI was a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
units on a scale | -5.8 (0.34) | -10.0 (0.5) | -10.7 (0.31)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -4.2, 95% CI 2-sided [-5.31 to -3.02] — Dupilumab 300 mg q2w v Placebo

18. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) to Week 16
Description: The POEM was a 7-item questionnaire that assessed disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
units on a scale | -5.3 (0.41) | -12.7 (0.64) | -12.9 (0.37)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -7.4, 95% CI 2-sided [-8.85 to -5.93] — Dupilumab 300 mg q2w v Placebo

19. Secondary Outcome: Change From Baseline in Hospital Anxiety Depression Scale (HADS) to Week 16
Description: HADS is a fourteen item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
units on a scale | -4.0 (0.37) | -4.9 (0.58) | -5.4 (0.35)
Statistical Analysis 1: Comparison: Placebo qw vs Dupilumab 300 mg q2w; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.1596, ANCOVA — Threshold for significance at 0.025 level; LS mean difference = -1.00, 95% CI 2-sided [-2.27 to 0.37] — Dupilumab 300 mg q2w v Placebo

20. Secondary Outcome: Percent Change From Baseline in Total Global Individual Signs Score (GISS) to Week 16
Description: Individual components of the AD lesions (erythema, infiltration/ papulation, excoriations, and lichenification) were rated globally (each assessed for the whole body, not by anatomical region) on a 4-point scale (0= none, 1= mild, 2= moderate and 3= severe) using the EASI severity grading criteria. Total score ranges from 0 (absent disease) to 12 (severe disease).
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percent change | -33.3 (1.89) | -55.4 (2.69) | -59.3 (1.64)

21. Secondary Outcome: Proportion of Topical Atopic Dermatitis Medication-Free Days Through Week 52
Description: Proportion of topical AD medication-free days through Week 52 was calculated as the number of days that a participant used neither topical corticosteroid (TCS)/ topical calcineurin inhibitors (TCI) nor system rescue therapy divided by the study days of each period.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
days | 10.5 (23.68) | 16.6 (30.08) | 22.5 (33.69)

22. Secondary Outcome: Percent Change From Baseline in Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score to Week 2
Description: as for outcome 7
Time Frame: Baseline to Week 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 106 | 319
percent change | -19.7 (1.58) | -27.3 (2.67) | -25.7 (1.57)

23. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score to Week 52
Description: as for outcome 14
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
percent change | -60.9 (4.29) | -84.9 (6.73) | -87.8 (6.19)

24. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Atopic Dermatitis to Week 52
Description: as for outcome 15
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percentage of BSA
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
Percentage of BSA | -29.41 (1.443) | -43.75 (1.874) | -43.67 (1.143)

25. Secondary Outcome: Percent Change From Baseline in the SCORing Atopic Dermatitis (SCORAD) Score to Week 52
Description: as for outcome 16
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
percent change | -47.3 (2.18) | -69.7 (3.06) | -70.4 (1.72)

26. Secondary Outcome: Percent Change From Baseline in Global Individual Signs Score (GISS) to Week 52
Description: as for outcome 20
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
percent change | -40.8 (2.72) | -62.8 (3.35) | -64.4 (2.13)

27. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) to Week 52
Description: as for outcome 17
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
units on a scale | -7.2 (0.4) | -11.4 (0.57) | -11.1 (0.36)

28. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) to Week 52
Description: The POEM was a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
units on a scale | -7.0 (0.57) | -14.2 (0.78) | -13.2 (0.45)

29. Secondary Outcome: Change From Baseline in Hospital Anxiety Depression Scale (HADS) to Week 52
Description: HADS is a fourteen item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire is scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
Time Frame: Baseline to Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 264 | 89 | 270
units on a scale | -3.8 (0.47) | -5.5 (0.71) | -5.9 (0.42)

30. Secondary Outcome: Number of Flares Through Week 52
Description: Atopic dermatitis (AD) flares were defined as worsening of the disease that required escalation/intensification of AD treatment. Number of flares occurred in the participants starting from first dose through Week 52 were reported.
Time Frame: Baseline up to Week 52
Population: All safety analysis were performed on safety analysis set (SAF) that included all randomized participants who received any study drug, and were analyzed as-treated.
Measure: Number; unit: flares
Groups:
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 51. During weeks in which Dupilumab was not administered, participants received placebo. Four participants received fewer injections of Dupilumab 300 mg in Dupilumab 300 qw arm, were analyzed in Dupilumab 300 mg q2w arm.
- Dupilumab 300 mg qw: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by a single 300 mg injection of Dupilumab qw from Week 1 to Week 51. Four participants received fewer injections of Dupilumab 300 mg in Dupilumab 300 qw arm, were analyzed in Dupilumab 300 mg q2w arm.
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
flares | 216 | 20 | 51

31. Secondary Outcome: Number of Serious Treatment Emergent Adverse Events (TEAEs) Leading to Study Drug Discontinuation Through Week 52
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. A Serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline up to Week 52
Population: All safety analysis were performed on SAF that included all randomized participants who received any study drug, and was analyzed as-treated.
Measure: Number; unit: events
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
events | 28 | 2 | 10

32. Secondary Outcome: Percentage of Participants With Skin Infection Treatment Emergent Adverse Events (TEAEs) (Excluding Herpetic Infections) From Baseline Through Week 52
Description: Any untoward medical occurrence in a participants who received IMP was considered an AE without regard to possibility of causal relationship with this treatment. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to end of treatment at Week 52). Any TEAE included participants with both serious and non-serious AEs. Skin infection TEAEs were identified based on blinded adjudication of all reported TEAEs under the 2 primary System Organ Classes (SOC): SOC = "Infection and Infestations" or SOC = "Skin and Subcutaneous Tissue Disorders". Blinded adjudication was performed and finalized by the study medical monitor before database lock.
Time Frame: Baseline up to Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
percentage of participants | 17.8 | 10.9 | 8.3

33. Secondary Outcome: Number of Skin Infection TEAEs (Excluding Herpetic Infections) From Baseline Through Week 52
Description: Any untoward medical occurrence in a participant who received IMP was considered an AE without regard to possibility of causal relationship with this treatment. TEAEs were defined as AEs that developed or worsened or became serious during on-treatment period (time from the first dose of study drug up to end of treatment at Week 52). Any TEAE included participants with both serious and non-serious AEs. Skin infection TEAEs were identified based on blinded adjudication of all reported TEAEs under the 2 primary System Organ Classes (SOC): SOC = "Infection and Infestations" or SOC = "Skin and Subcutaneous Tissue Disorders". Blinded adjudication was performed and finalized by the study medical monitor before database lock.
Time Frame: Baseline up to Week 52
Population: as for outcome 31
Measure: Number; unit: events
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
events | 80 | 15 | 29

34. Secondary Outcome: Percentage of Participants With Skin Infection Treatment Emergent Adverse Events (TEAEs) (Excluding Herpetic Infections) Requiring Systemic Treatment From Baseline Through Week 52
Description: as for outcome 33
Time Frame: Baseline up to Week 52
Population: as for outcome 31
Measure: Number; unit: percentage of participants
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
percentage of participants | 9.5 | 5.5 | 3.8

35. Secondary Outcome: Number of Skin Infection Treatment Emergent Adverse Events (TEAEs) (Excluding Herpetic Infections) Requiring Systemic Treatment From Baseline Through Week 52
Description: as for outcome 33
Time Frame: Baseline up to Week 52
Population: as for outcome 31
Measure: Number; unit: events
Groups:
- Dupilumab 300 mg q2w: Two subcutaneous injections of Dupilumab 300 mg (for a total of 600 mg) as a loading dose on Day 1, followed by placebo (for Dupilumab) alternating with single 300 mg injection of Dupilumab q2w from Week 1 to Week 51. During weeks in which Dupilumab was not administered, participants received placebo.Four participants received fewer injections of Dupilumab 300 mg in Dupilumab 300 qw arm, were analyzed in Dupilumab 300 mg q2w arm.
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 315 | 110 | 315
events | 44 | 7 | 13

36. Other Pre Specified Outcome: Change From Baseline in Sinonasal Outcome Test (SNOT-22) Score to Week 16
Description: The SNOT 22 was a validated measure of health related quality of life in sinonasal disease. It was a 22 item questionnaire with each item assigned a score ranging from 0-5. The total score may range from 0 (no disease) -110 (worst disease) (lower scores represent better health related quality of life). The SNOT-22 was administered only to participants with chronic inflammatory conditions of the nasal mucosa and/or paranasal sinuses.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 99 | 45 | 99
units on a scale | -4.77 (1.903) | -6.38 (2.445) | -10.39 (1.63)

37. Other Pre Specified Outcome: Change From Baseline in Asthma Control Questionnaire-5 (ACQ-5) Score to Week 16
Description: ACQ-5 questionnaire was a validated questionnaire comprising of 5 questions for asthma symptoms: woken at night by symptoms, wake in the mornings with symptoms, limitation of daily activities, shortness of breath, and wheeze. Participants were asked to rate their asthma symptoms during the previous week on a 7-point scale as 0=no impairment, 6=maximum impairment. ACQ-5 score was the mean of the 5 questions and range between 0 (totally controlled) and 6 (severely uncontrolled) (a higher score indicated lower asthma control). The ACQ-5 questionnaire was administered only to the participants with a medical history of asthma.
Time Frame: Baseline to Week 16
Population: All efficacy analyses were performed on the FAS, which included all randomized participants. Efficacy analyses were based on the treatment allocated by the IVRS/IWRS at randomization (as randomized). Here, number of participants analyzed = participants with ACQ-5 value at baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
Number analyzed (Participants) | 154 | 48 | 145
units on a scale | -0.12 (0.082) | -0.19 (0.113) | -0.36 (0.068)

ADVERSE EVENTS:
Time Frame: Time-frame was 'On treatment (Week 52) period' defined time from administration of first dose of study drug to study completion date of Week 52 visit (365 days starting from first dose of study drug if the date of Week 52 visit was unavailable).
Description: All Adverse Events (AEs) were collected from signature of informed consent form up to study completion date of the Week 52 visit regardless of seriousness or relationship to investigational product. Reported AEs and deaths are treatment-emergent that is AEs that developed/worsened and deaths that occurred during 'On treatment (Week 52) period'. Analysis was performed on SAF.
Arm/Group | Placebo qw | Dupilumab 300 mg q2w | Dupilumab 300 mg qw
All-Cause Mortality (participants affected / at risk) | 0/315 | 0/110 | 1/315
Serious Adverse Events (participants affected / at risk) | 20/315 | 4/110 | 12/315
Other Adverse Events (participants affected / at risk) | 216/315 | 74/110 | 228/315
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo qw (N=315) | Dupilumab 300 mg q2w (N=110) | Dupilumab 300 mg qw (N=315)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo qw (N=315) | Dupilumab 300 mg q2w (N=110) | Dupilumab 300 mg qw (N=315)
Blepharitis (Eye disorders) | 3 (3) | 6 (7) | 11 (14)
Conjunctivitis allergic (Eye disorders) | 19 (22) | 13 (20) | 54 (74)
Injection site reaction (General disorders) | 24 (102) | 16 (34) | 60 (224)
Influenza (Infections and infestations) | 17 (25) | 4 (4) | 9 (13)
Nasopharyngitis (Infections and infestations) | 62 (89) | 26 (40) | 63 (88)
Oral herpes (Infections and infestations) | 10 (15) | 4 (9) | 17 (31)
Sinusitis (Infections and infestations) | 9 (11) | 2 (2) | 18 (20)
Upper respiratory tract infection (Infections and infestations) | 34 (52) | 11 (21) | 46 (78)
Urinary tract infection (Infections and infestations) | 14 (16) | 2 (3) | 16 (22)
Headache (Nervous system disorders) | 19 (30) | 5 (5) | 24 (48)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 5 (5) | 7 (7)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 161 (278) | 40 (52) | 91 (133)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Not less than 45 days prior to submission for publication or presentation, the Institution shall, or cause the Principal Investigator to, provide the Sponsor with a copy of the Manuscript. The Institution shall consider in good faith any comments from the Sponsor regarding the content, and shall delete Confidential Information upon written request of the Sponsor. At the Sponsor's request, the Institution shall delay publication for an additional 60 days to allow patent applications to be filed.